CLINICAL TRIAL: NCT06543680
Title: Resin Modified Glass Ionomer Versus Self-Adhesive Resin Composite Restorative Systems: Two Years Randomized Clinical Study in Class ᴠ
Brief Title: Resin Modified Glass Ionomer Versus Self-Adhesive Resin Composite Restorative Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elbahloul, Assistant Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0103023CD
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Secondary Caries Dental Restoration Failure of Marginal Integrity

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be performed. A number of 35 patients will be included in this study. Each patient will have at least three NCCLs. One of these lesions will be randomly restored with resin modified glass ionomer cement, the second lesion will be restored with self-adhesive Surefil One composite hybrid while the third lesion will be restored with self-adhesive flowable composite.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resin Modified Glass Ionomer cement (Active Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Other: Dental restoration
- Self-Adhesive flowable composite (Placebo Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Other: Dental restoration
- Self-Adhesive composite hybrid (Placebo Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Other: Dental restoration

INTERVENTIONS:
Other: Dental restoration — Each patient will randomly receive one cervical restoration with one of the tested restorative systems

SUMMARY:
To evaluate and compare two-year clinical performance of commercially available resin modified glass ionomer cement, self-adhesive composite hybrid and self-adhesive flowable composite restorative materials for non-carious cervical lesions

DETAILED DESCRIPTION:
The experimental design description adhered to the guidelines provided by the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study is planned as a double-blinded randomized clinical trial, ensuring that both the patients and the examiner are unaware of the treatment allocation. The trial will follow a parallel design. A total of 35 patients, who are seeking dental treatment, will be enrolled in the study. The participants will be recruited from the Operative Department clinic at the Faculty of Dentistry, University of Mansoura. The study will focus on 105 Class V restorations.A randomized clinical trial will be performed. A number of 35 patients will be included in this study. Each patient will have at least three NCCLs. One of these lesions will be randomly restored with resin modified glass ionomer cement, the second lesion will be restored with self-adhesive Surefil One composite hybrid while the third lesion will be restored with self-adhesive flowable composite.

No active advertisement will be used for participant recruitment, and instead, a convenience sample will be formed. Prior to participating in the study, each patient will be required to provide informed consent by signing a consent form. The study is scheduled to be conducted from may 2023 to may 2025. The form and protocol of the study will be approved by Mansoura University's ethics committee before initiation.

Clinical evaluation for all restorations will be done at baseline (after insertion) and after 6, 12 and 24 months of clinical service by two calibrated independent examiners that will not share in restorations placement. It will be designed depending on modified USPHS criteria and FDI criteria

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be fair oral hygiene patients with 30-60 years. Patients with at least three similarly sized non-carious cervical lesions (NCCLs) in vital teeth that need for restoration and depth of NCCLs will be 1-3 mm with at least 50% of margins without enamel.

Exclusion Criteria:

* Exclusion criteria will be patients with severe periodontitis, mobile teeth, fractures, severe bruxism, carious teeth, poor oral hygiene, teeth with irreversible pulpitis and endodontically treated teeth.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-05-29 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of aesthetic, functional and biological properties for each group | 2 years after restoration
  Percentage of aesthetic, functional and biological properties that will be clinically assessed using World Dental Federation and USPHS parameters for each restorative system group

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Hamouda, Assistant Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Egypt
Locations (1):
- Faculty of dentistry mansoura university, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 Months for 2 years
Access Criteria: For any one